CLINICAL TRIAL: NCT00618501
Title: Gleevec (Imatinib) Plus Multi-Agent Chemotherapy For Newly-Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: Imatinib Mesylate and Combination Chemotherapy With or Without a Donor Stem Cell Transplant in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000586176; AMC-UUCM-2005-0238; NOVARTIS-AMC-UUCM-2005-0238
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2009-01

CONDITIONS: Leukemia
Keywords: untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cytarabine; Daunorubicin; Etoposide; Imatinib Mesylate; Leucovorin; Methotrexate; Prednisolone; Hydrocortisone; Vincristine

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: imatinib mesylate
Drug: leucovorin calcium
Drug: methotrexate
Drug: prednisolone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Imatinib mesylate may also stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known which treatment regimen is most effective in treating acute lymphoblastic leukemia.

PURPOSE: This phase II trial is studying the side effects of giving imatinib mesylate together with combination chemotherapy with or without a donor stem cell transplant and to see how well it works in treating patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the clinical efficacy of imatinib mesylate and combination chemotherapy in terms of complete response (CR) rate (both hematologic and molecular), CR duration, and overall survival in patients with newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia.
* To determine the toxicities of this regimen in these patients.

Secondary

* To establish the prognostic factors in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to age (64 or less vs 65 or over).

* Induction chemotherapy: Patients receive daunorubicin hydrochloride IV continuously over 24 hours on days 1-3, vincristine IV on days 1 and 8, and oral prednisolone on days 1-14. Treatment repeats for 5 courses in the absence of disease progression or unacceptable toxicity.
* Imatinib mesylate administration: Patients also receive oral imatinib mesylate once daily beginning on day 8 of course 1 induction chemotherapy and continuing for up to 2 years.
* Consolidation chemotherapy: Patients receive daunorubicin hydrochloride IV continuously over 24 hours on days 1-2, vincristine IV on days 1 and 8, and oral prednisolone on days 1-14 in course 1; cytarabine IV over 2 hours and etoposide IV over 3 hours on days 1-4 in courses 2 and 4; and methotrexate IV continuously over 36 hours on days 1-2 and 15-16 and leucovorin calcium IV every 6 hours x 3 doses followed by oral leucovorin calcium until methotrexate levels are < 0.05 micromol/L in courses 3 and 5. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with available HLA-matched sibling or unrelated hematopoietic cell donors or HLA-nonidentical familial hematopoietic cell donors proceed to allogeneic hematopoietic stem cell transplantation (HSCT). Patients who are without hematopoietic cell donors and who remain in hematologic remission continue to receive maintenance therapy with oral imatinib mesylate.
* Allogeneic HSCT: Patients undergo HSCT.
* CNS prophylaxis: Patients receive six doses of intrathecal (IT) methotrexate and hydrocortisone beginning on the first day of each chemotherapy course. Patients with CNS disease at diagnosis receive intensified CNS therapy comprising 10 doses of IT methotrexate and cranial irradiation after bone marrow remission is achieved.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute lymphoblastic leukemia (ALL) or acute mixed lineage leukemia

  * Newly diagnosed disease
  * Philadelphia-chromosome positive (Ph+) acute lymphoblastic leukemia or Ph+ acute mixed lineage leukemia

    * Positive result for RT-PCR for Bcr-Abl transcript (Ph+ ALL or Philadelphia-chromosome positive acute mixed lineage leukemia)

PATIENT CHARACTERISTICS:

* Bilirubin < 2 mg/dL
* SGOT < 3 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Ejection fraction > 45% by MUGA scan
* Not nursing
* Fertile patients must use effective contraception
* No known sensitivity to study drugs
* No severe medical conditions that, in the view of the investigator, prohibits participation in the study

PRIOR CONCURRENT THERAPY:

* No other investigational agents in the past 30 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving hematologic and molecular complete response (CR) after induction chemotherapy and imatinib mesylate
Duration of hematologic CR
Durations of hematologic and molecular CR after hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
Overall survival
Clinical toxicities
Prognostic factors in patients treated with this regimen

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea